CLINICAL TRIAL: NCT01352767
Title: A Randomised, Controlled, Cross-over Study With Inpatient and Outpatient Phases
Brief Title: The InsuPad in Daily Life Study - Effect of Local Heating on Postprandial Glucose Excursions Using the InsuPad Device
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insuline Medical Ltd. (Industry)
Collaborators: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-PP-002
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2012-05

CONDITIONS: Type 1 Diabetes Mellitus With Diabetic Neuralgia
Keywords: insulin injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- InsuPad Device (Experimental): Use of the InsuPad which heats the injection site.
  Interventions: Device: InsuPad
- CONTROL (No Intervention): no treatment

INTERVENTIONS:
Device: InsuPad — Heating pad
  Arms: InsuPad Device

SUMMARY:
A randomised, controlled, cross-over study with inpatient and outpatient phases. The inpatient phase length will be two days, which include a "Control" day without activating the InSuPad and a "Test" day where the InsuPad is activated. The outpatient phase length is 8 weeks: 4 weeks without the device-"Control", and 4 weeks with the device-"Test".

DETAILED DESCRIPTION:
A randomised, controlled, cross-over study with inpatient and outpatient phases. The inpatient phase length will be two days, which include a "Control" day without activating the InSuPad and a "Test" day where the InsuPad is activated. The outpatient phase length is 8 weeks: 4 weeks without the device-"Control", and 4 weeks with the device-"Test". Each subject will be randomly selected into one of two groups, group "A" and group "B". Forty (40) type I subjects who are meeting the inclusion/exclusion criteria as outlined below and who provide written Informed Consent will be enrolled in the study.

During the inpatient phase subjects will have standardized breakfast and dinner and venous blood samples will be taken for insulin and blood glucose measurements. Comparison of the two days ("control" and "test") will enable us to evaluate the effect of the device on post prandial glucose levels and insulin levels.

During the outpatient (daily life) phase subjects will be required to perform at least 5 self blood glucose measurements (SMBG), three before each meal and two at 90 minutes post breakfast and dinner. Comparing the SMBG measurement from the two periods will enable us to evaluate the effect of the device on post prandial glucose levels. The subjects will be contacted over the phone by the study staff to verify compliance with the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 70 years (values included)
* Type 1 diabetes mellitus or insulin treated type 2 diabetes with daily insulin demand ≥ 0.7 units per kg bodyweight.
* 6% ≤ HbA1c ≤ 9.5%
* Use of short-acting prandial insulin analogues with injections
* Study subject is willing to perform at least 5 blood glucose measurements per day for at least 56 days, willing to comply with study procedures and to keep a detailed patient log book.
* Willing to sign informed consent

Exclusion Criteria:

* Excessive fibrosis, lipo-hypertrophy or eczema at injection sites.
* Known gastro- or enteroparesis.
* Unstable chronic disease other than type 1 diabetes (e.g. Unstable angina factoris, , renal disease) for the last six months before study start.
* Severe hypoglycemic events requiring glucagon injection or glucose infusion within the last four weeks prior to study start.
* Hypoglycaemia unawareness (Score > 4 in the Hypoglycaemia Awareness Questionnaire, see appendix)
* Diabetic ketoacidosis (severe, with hospitalization) within the last six months prior to study start
* Any known life-threatening disease
* Pregnant women, lactating women or women who intend to become pregnant during the observation period
* Any other condition or compliance issues that might interfere with study participation or results
* Subjects with heat sensitivity
* Subjects involved in or planed to participate in other studies
* Subjects who are incapable of contracting or under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
efficacy | 2 hours
  AUC120 BG (area under the curve of postprandial glucose change 2 hours after meal) after breakfast and dinner under standardized conditions during the inpatient phase.

SECONDARY OUTCOMES:
Efficacy | 8 weeks
  Mean change in post prandial glucose level at 90 minutes during the outpatient phase.
Efficacy | 8 weeks
  AUC60 Ins (area under the curve of insulin concentration change 1 hour after meal) after breakfast and dinner under standardized conditions during the inpatient phase.
Safety | 14 weeks
  • Number and severity of hypoglycaemias and hyperglycaemias and assessment of relationship to the use of the InsuPad device during the whole study.
Satisfaction | 14 weeks
  • Patient satisfaction (subjective clinical performance) at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Bad Mergentheim, Bad Mergentheim, Germany

REFERENCES:
- See also: Related Info — http://www.insuline-medical.com